CLINICAL TRIAL: NCT01962064
Title: Social Cognition in Ageing and in Frontotemporal Lobar Degeneration (Frontotemporal Dementia and Semantic Dementia): a Cognitive and Neuroimaging Study
Brief Title: Social Cognition in Ageing and in Frontotemporal Lobar Degeneration
Acronym: COSIMAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-A00681-40
Record Dates: First submitted 2013-09-03; First posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Frontotemporal Lobar Degeneration; Aging
MeSH Terms: conditions — Frontotemporal Lobar Degeneration | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Semantic demantia (Experimental): cognitive assessment and Brain imaging examination MRI of patient with the semantic variant of primary progressive aphasia
  Interventions: Behavioral: Cognitive assessment; Other: Brain imaging examination MRI
- Frontotemporal dementia (Experimental): cognitive assessment and Brain imaging examination MRI of patients with the behavioral variant of frontotemporal lobar degeneration
  Interventions: Behavioral: Cognitive assessment; Other: Brain imaging examination MRI
- Elderly (Experimental): cognitive assessment and Brain imaging examination MRI of healthy elderly subjects
  Interventions: Behavioral: Cognitive assessment; Other: Brain imaging examination MRI
- Young (Experimental): cognitive assessment and Brain imaging examination MRI of young subjects
  Interventions: Behavioral: Cognitive assessment; Other: Brain imaging examination MRI

INTERVENTIONS:
Behavioral: Cognitive assessment
Other: Brain imaging examination MRI

SUMMARY:
The purpose of this study is to examine the age and the neurodegenerative disease effects on social cognition. Secondary goals are to better understand the relationships between different component of social cognition, executive functioning, and behavior and describing the neuronal substrates associated to the alteration of the social cognition in ageing and dementia.

ELIGIBILITY:
Inclusion Criteria:

* All the participants

  * Age between 40 and 80 years
  * Minimum of 7 years of education
  * French native speaker
* Healthy subjects

  * Non pathological Dementia rating scale score
* Patients

  * Clinical diagnosis of frontotemporal lobar degeneration

Exclusion Criteria:

* Chronic neurological disease
* Encephalitis
* Endocrinal disease
* Hepatic disease
* Case history of head injury with loss of consciousness of more than one hour
* Case history of stroke
* Case history of cancer during the five last years except squamous cell carcinomas
* Alcoholism or drug addiction
* Major psychiatric disorders according the Diagnostic and Statistical Manual of Mental Disorders

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-07 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Social cognition scores | 2 years
  number of correct responses in a social cognition test

CONTACTS AND LOCATIONS:
Overall Officials: Vincent de La Sayette, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- Inserm - EPHE - University of Caen U1077, Caen, France